CLINICAL TRIAL: NCT05161338
Title: Impact of Vaginal Microbiome on Vaginal Absorption of Exogenous Progesterone: a Pilot Study.
Acronym: PROGEBIOMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2110-VLC-095-EL
Record Dates: First submitted 2021-12-15; First posted 2021-12-17 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Infertility, Female
Keywords: LUTHEAL PHASE SUPPORT; MICROBIOME; INFERTILITY; ONGOING PREGNANCY RATE; LIFE BIRTH RATE; ARTIFICIAL REPRODUCTION TREATMENT; EMBRYO TRANSFER
MeSH Terms: conditions — Infertility, Female; Infertility

STUDY DESIGN:
Intervention Model Description: Prospective cohort unicentric pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FROZEN EMBRYO TRANSFER (Experimental): Women who undergo an artificial cycle for frozen embryo transfer and receive luteal phase support.
  Interventions: Diagnostic Test: MICROBIOME GENETIC ANALYSIS; Diagnostic Test: VAGINAL PH VALUE; Diagnostic Test: SERUM PROGESTERONE LEVELS; Diagnostic Test: SERUM OESTRADIOL LEVELS

INTERVENTIONS:
Diagnostic Test: MICROBIOME GENETIC ANALYSIS — Vaginal samples will be taken. A floxed nylon swab will be rotated against the posterior vaginal wall, Nucleic acid extraction and genetic analisys will be performed
Diagnostic Test: VAGINAL PH VALUE — Intravaginal Ph value meassurement.
Diagnostic Test: SERUM PROGESTERONE LEVELS — Determination of serum P4 levels On the day of embryo transfer scheduling (prior to the onset of exogenous progesterone administration) and on the embryo transfer day-.
Diagnostic Test: SERUM OESTRADIOL LEVELS — Determination of serum E2 levels On the day of embryo transfer scheduling (prior to the onset of exogenous progesterone administration) and on the embryo transfer day.

SUMMARY:
Is already demonstrated that around 30% of patients undergoing an artificial cycle with vaginal progesterone do not reach a minimum threshold value of serum progesterone levels on the day of embryo transfer. Women with serum progesterone levels below this threshold have 20% lower ongoing pregnancy and live birth rates, decreasing their chances of success. However, the cause of this high heterogeneity in exogenous vaginal progesterone absorption among our patients remains unknown. It has been suggested that vaginal microbiome, and vaginal pH (due to its impact in microbiota growth), may explain the differences in vaginal progesterone absorption. The aim of the present pilot study is to assess if certain vaginal conditions, such as its microbiome status or its pH level, might affect vaginal progesterone absorption (measured by serum progesterone levels) and, in turn, the chances of success. In order to evaluate it, a prospective cohort unicentric study will be conducted in IVI RMA Valencia (Spain). Infertile patients undergoing an embryo transfer in the context of an artificial cycle when using vaginal progesterone will be recruited. Serum progesterone and estradiol levels, microbiome genetic analysis in vaginal samples and vaginal pH will be measured both on the embryo transfer-scheduling day and on the embryo transfer day.

DETAILED DESCRIPTION:
Currently, as part of routine clinical practice serum progesterone levels were meassured of women undergoing an ET in the context of an artificial cycle. These blood tests are usually performed around 2 hours before ET, thus results are available before their departure of the clinic. In the event of detecting low serum progesterone levels, an extra dose of exogenous subcutaneous progesterone is given for LPS.

There is not knowing about the reason of this heterogeneity in progesterone absorption, and one plausible hypothesis is vaginal microbiome. In the event of proving a significant association between vaginal microbiome and serum progesterone levels on the day of ET, and in particular if these levels are below or above the delimited threshold, it would be possible to individualize LPS in several patients in a more direct manner.

It is true that our current clinical practice, giving subcutaneous progesterone, is capable of equaling OPR of women with serum progesterone levels below 8.8 ng/ml on the ET day to those with values above this threshold applying the exact same approach to all patients. This study could be the next step towards an iLPS, to know the reason of the lower progesterone levels, and treat it directly, instead of moving to the need of a daily injection of progesterone which is costly and not patient friendly. Furthermore, vaginal microbiome may also have an impact in the subsequent OPR, even though serum progesterone levels were over 8.8 ng/ml. If this is the case, the analisys in advance the patient's vaginal microbiome will allow to treat the patient accordingly in order to increase the results of the ART treatment.

ELIGIBILITY:
Inclusion Criteria:

* The subject must provide written informed consent prior to any study related procedures
* Women ≤50 years old
* BMI ≤ 25 kg/m2
* Adequate endometrial thickness (>6.5mm) and pattern (Triple A structure) in the proliferative phase

Exclusion Criteria:

* Uterine Pathology, adnexal pathology
* Systemic diseases -

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Vaginal Microbiome | 12 months
  Result of the microbiome genetic analysis in vaginal samples (nucleic acid extraction and genetic analysis)

SECONDARY OUTCOMES:
Live birth | 12 months
  Live birth rate
Ongoing Pregnancy Rate | 12 months
  Success value in pregnancy after ultrasound confirmation of heartbeat and 12 weeks of pregnancy
Clinical Pregnancy | 12 months
  Pregnancy confirmation by the observation of the presence of at least one gestational sac on ultrasound
Serum progesterone value | 12 months
  Serum progesterone levels
Vaginal PH | 12 months
  Measure of vaginal pH levels

CONTACTS AND LOCATIONS:
Locations (1):
- Ivi Valencia, Valencia, Spain